CLINICAL TRIAL: NCT05046665
Title: A Single-centre, Open-label, Phase I Study to Evaluate the Diagnostic Performance of 89Zirconium-labelled Girentuximab (89Zr-TLX250) PET in Urothelial Cancer Patients (ZiPUP Study)
Brief Title: Phase I Study to Evaluate the Diagnostic Performance of 89Zirconium Girentuximab PET in Urothelial Cancer Patients
Acronym: ZiPUP
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: South Metropolitan Health Service (Other Government)
Collaborators: Telix Pharmaceuticals (Innovations) Pty Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ZiPUP; NCT05018442 (obsolete NCT alias)
Record Dates: First submitted 2021-09-08; First posted 2021-09-16 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Urothelial Carcinoma
Keywords: Glandular and Epithelial
MeSH Terms: conditions — Carcinoma, Transitional Cell

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Administration of 89Zr-Girentuximab (Other): Administration of 89Zr-Girentuximab as per protocol
  Interventions: Drug: 89Zr-Girentuximab

INTERVENTIONS:
Drug: 89Zr-Girentuximab — Administration of 89Zr-girentuximab as per protocol.

SUMMARY:
The aim of this study is to determine if it is practical to use 89Zr-TLX250 PET/CT in the staging and detection of localized and metastatic urothelial carcinoma or bladder cancer.

The primary objective is to evaluate the feasibility of using 89Zr-TLX250 PET/CTas a new diagnostic and staging modality to detect urothelial carcinoma or bladder cancer.

DETAILED DESCRIPTION:
This will be a non-randomised, non-blinded, single centre, phase 1 feasibility study comparing 89Zr-girentuximab PET with FDG PET in patients with urothelial carcinoma or bladder cancer. This study would include 2 cohorts of adult patients; those with known metastatic urothelial carcinoma and bladder cancer and those undergoing primary staging for recently diagnosed urothelial carcinoma or bladder cancer.

This study is open-label, single centre and eligible patients will receive a single administration of study drug prior to imaging on day 5 (+/- 2 days). PET scans will be independently interpreted by nuclear medicine physicians blinded to the FDG PET findings. For patients proceeding to radical cystectomy, subsequent histological confirmation of areas of increased uptake will be retrospectively correlated with both PET scans.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 or older with bladder cancer or urothelial carcinoma who are able to provide informed consent
2. Negative serum pregnancy test in female patients of childbearing potential at screening. Confirmation of negative pregnancy test result from urine within 24 hours prior to receiving investigational product.
3. Consent to practise double-barrier contraception until a minimum of 42 days after 89Zr-TLX250 administration.

Exclusion Criteria:

1. Active malignancy other than urothelial carcinoma or bladder cancer
2. Administration of a radioisotope within 10 physical half-lives prior to study enrolment.
3. Administration of chemotherapy, radiotherapy, or immunotherapy within 4 weeks prior to planned administration of 89Zr-TLX250 or continuing adverse effects from such therapy
4. Planned antineoplastic therapies for the period between administration of 89Zr-TLX250 and imaging
5. Serious non-malignant disease that may interfere with the objectives of the study
6. Renal insufficiency with glomerular filtration rate ≤45 mL/min/1.73m2
7. Pregnancy or lactation
8. Exposure to murine or chimeric antibodies within the last 5 years
9. Known hypersensitivity or human anti-chimeric antibodies against girentuximab
10. Exposure to any experimental diagnostic or therapeutic drug 30 days prior to the date of planned administration of 89Zr-TLX250
11. Contraindications to FDG PET/CT

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2021-05-14 (Actual); Primary Completion 2022-08-09 (Actual); Study Completion 2022-08-09 (Actual)

PRIMARY OUTCOMES:
Comparison of the sensitivity and specificity of 89Zr-girentuximab PET with FDG PET | Day 1 - Day 90
  Sensitivity and specificity will be established following histological confirmation

SECONDARY OUTCOMES:
To evaluate the correlation between 89Zr-girentuximab SUV's and degree of urinary carbonic anhydrase IX excretion (cytology and CA-IX via PCR). | Day 1
  89Zr-girentuximab SUV's will be correlated with urinary CA-IX expression
Number of participants with treatment related adverse events related to 89Zr-girentuximab administration | Day 1 to Day 90
  Number of participants with treatment-related adverse events as assessed by NCI-CTCAE v 5.0 criteria
To quantify the correlation between tumour volume using MIM quantitative software and histopathological findings | Day 1 - Day 90
  Tumour burden as defined by volumetric software will be correlated with histopathological results

CONTACTS AND LOCATIONS:
Locations (1):
- Fiona Stanley Hospital, Murdoch, Western Australia, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Al-Zubaidi M, Viswambaram P, McCombie S, Liow E, Lenzo N, Ferguson T, Redfern AD, Gauci R, Hayne D. 89Zirconium-labelled girentuximab (89Zr-TLX250) PET in Urothelial Cancer Patients (ZiPUP): protocol for a phase I trial of a novel staging modality for urothelial carcinoma. BMJ Open. 2022 Apr 15;12(4):e060478. doi: 10.1136/bmjopen-2021-060478. PMID 35428649